CLINICAL TRIAL: NCT06377982
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Clinical Study to Assess the Safety and Efficacy of Allogeneic Human Umbilical Cord Blood Infusion in Children with Cerebral Palsy
Brief Title: Human Umbilical Cord Blood Infusion in Patients with Cerebral Palsy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: StemCyte Taiwan Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: StemCyte International, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCCP001
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hUCB treatment (Experimental): Human cord blood infusion
  Interventions: Biological: hUCB
- Placebo treatment (No Intervention): Placebo infusion

INTERVENTIONS:
Biological: hUCB — hUCB
  Arms: hUCB treatment

SUMMARY:
A phase I, randomized, double-blind, placebo-controlled clinical study to assess the safety and efficacy of allogeneic human umbilical cord blood infusion in children with cerebral palsy

DETAILED DESCRIPTION:
This is a phase I study to evaluate the safety and efficacy in hUCB treatment on the patients with cerebral palsy (CP).

ELIGIBILITY:
Inclusion Criteria:

* Male or female underage at the time of screening.
* With a confirmed diagnosis of CP
* non-progressive motor disability
* brain dysfunction

Exclusion Criteria:

* Judged by the Investigator to be not suitable/eligible for study participation.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
safety-TEAE | From screening to 56 weeks
  Frequency and incidence of treatment-emergent adverse events (TEAEs).

IPD SHARING:
Plan to Share IPD: No